CLINICAL TRIAL: NCT04499807
Title: Accuracy of Rhythm Detection and Managing Data Deluge by a Wearable Smart Watch for Cardiac Arrhythmias (The WATCH-RHYTHM Study)
Brief Title: Accuracy of Rhythm Detection by a Wearable Smart Watch for Cardiac Arrhythmias (The WATCH-RHYTHM Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped because after we started enrolling we realized that we could not get the information that we wanted out of the current protocol. The information we wanted to compare would not be able to be collected.
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KCHRF-WATCH RHYTHM-0006
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: Wearable technology; Smart Watch; ILR; AFib detection
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart Watch (Other): The patients will wear the Smart Watch to generate data to assess their rhythm as confirmed by the ILR done during the same time.
  Interventions: Other: AFib detection with wearable smart watch

INTERVENTIONS:
Other: AFib detection with wearable smart watch — Patients will transmit two rhythm strips every day through both the devices and additional transmission whenever they have symptoms (palpitations, skipped beats, shortness of breath and chest pain). The transmitted rhythm strips are de-identified and analyzed after assigning a unique ID for research purposes.

SUMMARY:
It is an attempt to see the reliability of the Wearable Smart Watch in identifying atrial fibrillation and other arrhythmias compared to the data detected from ILRs.

DETAILED DESCRIPTION:
The sensitivity, specificity, positive and negative predictive values for successful identification of normal sinus rhythm, atrial fibrillation and other rhythm disorders from the smart watch will compared to that of an ILR.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patients who have an implantable loop recorder for heart rhythm monitoring purposes
* Having IOS iphone device that can be integrated into Apple Watch
* Willing to sign a consent form and participate in the study

Exclusion Criteria:

* Hemodynamically unstable patients
* Over 90 years of age
* Presence of wrist tattoos
* Presence of AV fistula on the wrist on which the wearable is worn. (If the contralateral wrist is unaffected, those patients can be included)
* Presence of Implantable Cardiac Pacemaker and/or ICD
* Patients with Parkinsons disease or tremors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
AFib detection with heart rate data measured by Smart Watch | 5 months
  Heart rate data generated by Smart Watch is used to assess their rhythm as confirmed by the ILR done during the same time.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naccarelli GV, Varker H, Lin J, Schulman KL. Increasing prevalence of atrial fibrillation and flutter in the United States. Am J Cardiol. 2009 Dec 1;104(11):1534-9. doi: 10.1016/j.amjcard.2009.07.022. PMID 19932788
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Savelieva I, Camm J. Update on atrial fibrillation: part II. Clin Cardiol. 2008 Mar;31(3):102-8. doi: 10.1002/clc.20136. PMID 18383050
- [Background] Glotzer TV, Daoud EG, Wyse DG, Singer DE, Ezekowitz MD, Hilker C, Miller C, Qi D, Ziegler PD. The relationship between daily atrial tachyarrhythmia burden from implantable device diagnostics and stroke risk: the TRENDS study. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):474-80. doi: 10.1161/CIRCEP.109.849638. Epub 2009 Aug 4. PMID 19843914
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Mairesse GH, Moran P, Van Gelder IC, Elsner C, Rosenqvist M, Mant J, Banerjee A, Gorenek B, Brachmann J, Varma N, Glotz de Lima G, Kalman J, Claes N, Lobban T, Lane D, Lip GYH, Boriani G; ESC Scientific Document Group. Screening for atrial fibrillation: a European Heart Rhythm Association (EHRA) consensus document endorsed by the Heart Rhythm Society (HRS), Asia Pacific Heart Rhythm Society (APHRS), and Sociedad Latinoamericana de Estimulacion Cardiaca y Electrofisiologia (SOLAECE). Europace. 2017 Oct 1;19(10):1589-1623. doi: 10.1093/europace/eux177. No abstract available. PMID 29048522
- [Background] Stott DJ, Dewar RI, Garratt CJ, Griffith KE, Harding NJ, James MA, Lane DA, Petty DR, Smith PA, Somerville MH, Trueland J. RCPE UK Consensus Conference on 'approaching the comprehensive management of atrial fibrillation: evolution or revolution?'. J R Coll Physicians Edinb. 2012 Mar;42(1):34-5. doi: 10.4997/JRCPE.2012.S01. No abstract available. PMID 22441062
- [Background] Verkruysse W, Svaasand LO, Nelson JS. Remote plethysmographic imaging using ambient light. Opt Express. 2008 Dec 22;16(26):21434-45. doi: 10.1364/oe.16.021434. PMID 19104573
- [Background] McMANUS DD, Chong JW, Soni A, Saczynski JS, Esa N, Napolitano C, Darling CE, Boyer E, Rosen RK, Floyd KC, Chon KH. PULSE-SMART: Pulse-Based Arrhythmia Discrimination Using a Novel Smartphone Application. J Cardiovasc Electrophysiol. 2016 Jan;27(1):51-7. doi: 10.1111/jce.12842. Epub 2015 Nov 13. PMID 26391728
- [Background] McManus DD, Lee J, Maitas O, Esa N, Pidikiti R, Carlucci A, Harrington J, Mick E, Chon KH. A novel application for the detection of an irregular pulse using an iPhone 4S in patients with atrial fibrillation. Heart Rhythm. 2013 Mar;10(3):315-9. doi: 10.1016/j.hrthm.2012.12.001. Epub 2012 Dec 6. PMID 23220686
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- See also: Enforcement Policy for Non-Invasive Remote Monitoring Devices Used to Support Patient Monitoring During the Coronavirus Disease 2019 (COVID-19) Public Health Emergency (Revised) — https://www.fda.gov/media/136290/download